CLINICAL TRIAL: NCT06055205
Title: A Pain and Coordination Plan (PAC-plan) in Transition Between Hospital and Primary Care to Reduce Opioid Use in Patients After Accidental Injuries: A Randomized Controlled Trial
Brief Title: A Pain and Coordination Plan for Reduced Opioid Use After Accidental Injuries
Acronym: PAC-plan
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Oslo University Hospital (Other); The Norwegian Research Fund for General Practice (Unknown)
Responsible Party: Principal Investigator, Trygve Skonnord, Associate professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 487948 (REK)
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Opioid Use; Injury Traumatic; Pain, Postoperative
Keywords: Opioids; Injuries; Pain; Pain management; Collaboration
MeSH Terms: conditions — Wounds and Injuries; Pain, Postoperative; Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: The study will use a prospective randomized controlled trial design. Participants will be assigned randomly to study conditions (1:1) through permuted block randomization with various sizes of the blocks (4, 6, 8, 10) in random order. The randomization will be performed manually by the principle investigator (PI). Sealed, opaque, numbered envelopes will be used, and will be opened after consent from the patient. For the intervention group, the study coordinator will contact the patient's general practitioner (GP) by calling the doctor's office to obtain consent for participation. For the control group, the GP will not be asked for consent. To ensure that no GPs are included in both groups, the GPs retain their initial allocation if they have additional patients in the project. In practice, this corresponds to cluster-randomization at the GP level (and will be treated as such in the statistical analyzes).
Who Masked: Outcomes Assessor
Masking Description: The statistician performing the data analyses will be masked for group status. The participants, study nurses and study coordinator will not be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAC-plan (Experimental): The patients receive a Pain- and Coordination plan (PAC-plan) at discharge from the hospital. The PAC-plan includes:
  * Upon discharge, patients have a patient-centered conversation and receive written information covering patient education on opioids, a tapering plan, and a plan for contact and follow-up with the general practitioner. The information is based on the Norwegian National Guide for Addictive Medications.
  * Before discharge, patients are scheduled an appointment with the GP, preferably within the first 2 weeks (2-4 weeks), for a follow-up regarding the injury and pain management.
  * The GP is invited to maintain contact with the study nurse at the hospital for one year. The general practitioner can call for consultation with the study nurse, and if necessary, be connected with relevant medical specialists for advice and eventually further follow-up.
  Interventions: Other: PAC-plan
- Control (No Intervention): Treatment and follow-up as usual.

INTERVENTIONS:
Other: PAC-plan — The participants will be asked to complete electronic questionnaires at baseline, and at 6 weeks and 52 weeks after discharge from the hospital. The completion of these questionnaires will take place during the 6-week follow-up appointment at the hospital (a standard follow-up for all patients undergoing surgery at the Division of Orthopedic Surgery, Oslo University Hospital, Norway). Additionally, participants will be invited for a phone-based follow-up appointment with the study coordinator 52 weeks after discharge. The participants will receive the questionnaires electronically via SMS or email. If electronic options are not feasible, data can be collected through paper questionnaires sent by mail. Data will not be directly obtained from general practitioners.
  Arms: PAC-plan

SUMMARY:
This clinical trial aims to lower the number of people who use opioids and improve the quality of health in patients who have experienced accidental injury by implementing a Pain and Coordination Plan (PAC-plan). The PAC-plan will be given upon discharge from the hospital.

The main questions this study aims to answer are:

* Can the PAC-plan reduce opioid use in patients after accidental injuries?
* Can the PAC-plan increase quality of life in patients after accidental injuries?

Participants will be randomly assigned to the PAC-plan or usual care. The PAC-plan includes:

* an opioid management plan upon discharge from the hospital
* an appointment with his/her general practitioner within 2-4 weeks after discharge
* the general practitioner will be given the opportunity for increased collaboration with the hospital specialists

Participants in both groups will be asked to answer questionnaires about their health at discharge, and at 6 and 52 weeks after discharge from the hospital. In addition, the researchers will use data from the Norwegian Prescription Database to measure opioid use.

DETAILED DESCRIPTION:
Introduction: Patients experiencing serious injuries are at risk of developing long-term opioid use, yet many don't receive plans for opioid reduction when discharged from the hospital. General Practitioners (GPs) also experience insufficient communication from the hospital on pain management plans. Opioids are often essential for managing acute pain in patients following serious injuries. However, it is crucial to prioritize safe and appropriate pain management in subsequent phases. The opioid epidemic in the USA, characterized by opioid use disorders and addiction, has resulted in high mortality rates and a public health crisis. In 2017, opioid dependence outside the USA was estimated to account for over 1% of age-standardized years lived with disability in 135 countries. Considering the devastating impact of the opioid epidemic in the USA, it is imperative to draw lessons from these experiences and implement preventive measures to avoid a similar crisis in other countries.

Aim: This study aims to explore if a Pain and Coordination Plan (PAC-plan) for patients after accidental injury can reduce opioid use and improve quality of life.

Methods: The study is designed as a prospective randomized controlled trial (RCT) to evaluate the effect of a PAC-plan. The PAC-plan consists of three main elements: an opioid management plan upon discharge from the hospital, an appointment with the participant's regular GP within 2-4 weeks after discharge and an opportunity for increased collaboration between GP and hospital specialists.

Patients will be recruited from the Division of orthopaedic surgery, Oslo University Hospital (OUH), Norway. OUH is a highly specialized hospital in charge of extensive regional and local hospital assignments in the South-Eastern Health region in Norway and is described as a level 1 trauma centre. The primary outcome is oral morphine equivalent (OMEQ) consumption 6 weeks after discharge. Secondary outcome measures are OMEQ 52 weeks after discharge. In addition, registry-based OMEQ, pain, health-related quality of life (HRQoL) and other Patient-reported outcome measures (PROMs) at 6 and 52 weeks. The registry-based OMEQ will be collected from the Norwegian Prescription Database (NorPD). Data will also be collected from the the Norwegian Patient Registry (NPR).

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age who have undergone acute orthopaedic surgery following accidental injury
* Discharged on opioid medication

Exclusion Criteria:

* Unable to read, speak, and write Norwegian
* Severe cognitive impairment/inability to consent
* Not discharged to home
* Currently in cancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2023-09-25 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Opioid use | 6 weeks post-discharge
  Opioid use last 24 hours measured in oral morphine equivalents (OMEQ), self-reported

SECONDARY OUTCOMES:
Opioid use | 52 weeks post-discharge
  Opioid use last 24 hours measured in oral morphine equivalents (OMEQ), self-reported
Opioid use measured in oral morphine equivalents (OMEQ), registry-based | 6 weeks post-discharge
  The Norwegian Prescription Database, NorPD
Opioid use measured in oral morphine equivalents (OMEQ), registry-based | 52 weeks post-discharge
  The Norwegian Prescription Database, NorPD
Numeric Rating Scale for pain intensity scores | 6 weeks post-discharge
  Pain intensity, self-reported by Numeric Rating Scale (NRS-11). Scale from 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable."
Numeric Rating Scale for pain intensity scores | 52 weeks post-discharge
  Pain intensity, self-reported by Numeric Rating Scale (NRS-11). Scale from 0 to 10, with 0 being "no pain" and 10 being "the worst pain imaginable."
EQ-5D-5L (EuroQol, 5 dimensions, 5 levels) for health-related quality of life | 6 weeks post-discharge
  Health-related quality of life measured with the EQ-5D-5L. The EQ-5D-5L consists of two parts: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ visual analogue scale (EQ VAS) records the patient's self-rated health on a VAS ranging from 0 to 100, with higher scores indicating better self-reported health.
EQ-5D-5L (EuroQol, 5 dimensions, 5 levels) for health-related quality of life | 52 weeks post-discharge
  Health-related quality of life measured with the EQ-5D-5L. The EQ-5D-5L consists of two parts: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ visual analogue scale (EQ VAS) records the patient's self-rated health on a VAS ranging from 0 to 100, with higher scores indicating better self-reported health.
Norwegian Injustice Experience Questionnaire (IEQ-N) | 6 weeks post-discharge
  Perceived injustice measured with the Injustice Experience Questionnaire (IEQ). The IEQ is a self-report 12-item questionnaire and each item is scored on a five-point scale from zero ("never") to four ("all the time"). The total score on the IEQ ranges from 0 to 48, with higher scores indicating higher levels of perceived injustice
Norwegian Injustice Experience Questionnaire (IEQ-N) | 52 weeks post-discharge
  Perceived injustice measured with the Injustice Experience Questionnaire (IEQ). The IEQ is a self-report 12-item questionnaire and each item is scored on a five-point scale from zero ("never") to four ("all the time"). The total score on the IEQ ranges from 0 to 48, with higher scores indicating higher levels of perceived injustice
Life Orientation Test Revised (LOT-R) | 6 weeks post-discharge
  Optimism measured with the Life Orientation Test Revised (LOT-R). The measure consists of 10 items, and participants indicate their level of agreement with each item on a 5-point scale ranging from 0 (strongly disagree) to 4 (strongly agree). The scores on this scale can range from 0 to 24, with higher scores indicating greater levels of optimism and lower scores indicating lower levels of optimism.
Life Orientation Test Revised (LOT-R) | 52 weeks post-discharge
  Optimism measured with the Life Orientation Test Revised (LOT-R). The measure consists of 10 items, and participants indicate their level of agreement with each item on a 5-point scale ranging from 0 (strongly disagree) to 4 (strongly agree). The scores on this scale can range from 0 to 24, with higher scores indicating greater levels of optimism and lower scores indicating lower levels of optimism.
Patient Health Questionnaire-9 | 6 weeks post-discharge
  Depression symptoms and severity measured by the Patient Health Questionnaire-9 (PHQ-9).The PHQ-9 consists of nine items and the participants rate the frequency of each symptom on a Likert scale ranging from 0 (not at all) to 3 (nearly every day). The scores can range from 0-27. In addition to a total score, categories are defined to indicate severity of depression symptoms. These categories are defined as follows: none (total score from 0 to 4), mild (total score from 5 to 9), moderate (total score from 10 to 14), moderately severe (total score from 15 to 19), and severe (total score from 20 to 27).
Patient Health Questionnaire-9 | 52 weeks post-discharge
  Depression symptoms and severity measured by the Patient Health Questionnaire-9 (PHQ-9).The PHQ-9 consists of nine items and the participants rate the frequency of each symptom on a Likert scale ranging from 0 (not at all) to 3 (nearly every day). The scores can range from 0-27. In addition to a total score, categories are defined to indicate severity of depression symptoms. These categories are defined as follows: none (total score from 0 to 4), mild (total score from 5 to 9), moderate (total score from 10 to 14), moderately severe (total score from 15 to 19), and severe (total score from 20 to 27).
HUNT (the Nord-Trøndelag health study) physical activity questionnaire (HUNT 1 PA-Q) | 6 weeks post-discharge
  The HUNT 1 PA-Q consists of three sets of questions addressing the average number of times exercising each week, the average intensity and average hours each time. Each set of questions has five, three, or four response choices, respectively. The HUNT 1 PA-Q measures physical exercise as the product of average frequency (0.0-5.0 points), duration (0.10-1.00 points) and intensity (1-3 points) each week, giving an index ranging from 0.00 to 15.00, with 15.00 as the best score
HUNT (the Nord-Trøndelag health study) physical activity questionnaire (HUNT1 PA-Q) | 52 weeks post-discharge
  The HUNT 1 PA-Q consists of three sets of questions addressing the average number of times exercising each week, the average intensity and average hours each time. Each set of questions has five, three, or four response choices, respectively. The HUNT 1 PA-Q measures physical exercise as the product of average frequency (0.0-5.0 points), duration (0.10-1.00 points) and intensity (1-3 points) each week, giving an index ranging from 0.00 to 15.00, with 15.00 as the best score.
Insomnia Severity Index (ISI) last 2 weeks | 6 weeks post-discharge
  Perceived insomnia severity measured by the Insomnia Severity Index (ISI). The ISI consists of seven items and the participants rate each item on a scale from 0 to 4, from less to more severe. The total score is the sum of each individual item and can range from 0 to 28 (28 = most severe insomnia).
Insomnia Severity Index (ISI) last 2 weeks | 52 weeks post-discharge
  Perceived insomnia severity measured by the Insomnia Severity Index (ISI). The ISI consists of seven items and the participants rate each item on a scale from 0 to 4, from less to more severe. The total score is the sum of each individual item and can range from 0 to 28 (28 = most severe insomnia).

CONTACTS AND LOCATIONS:
Overall Officials: Lene B Solberg, PhD MD, Study Director — Oslo University Hospital; Trygve Skonnord, PhD MD, Principal Investigator — Department of General Practice, Institute of Health and Society, University of Oslo, Norway
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make individual patient data (IPD) available.

REFERENCES:
- See also: Website for the PAC-plan project at the University of Oslo — https://www.med.uio.no/helsam/english/research/projects/pain-and-coordination-plan/index.html